CLINICAL TRIAL: NCT03013517
Title: Open-label Follow-up Study of the PEPITES Study to Evaluate the Long-term Efficacy and Safety of Viaskin Peanut
Brief Title: Follow-up of the PEPITES Study to Evaluate Long-term Efficacy and Safety of Viaskin Peanut in Children
Acronym: PEOPLE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: DBV Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEOPLE
Expanded Access: NCT04371627 (No longer available)
Record Dates: First submitted 2017-01-02; First posted 2017-01-06 (Estimated); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Peanut Allergy
Keywords: Allergy; food allergy; viaskin; peanut; epicutaneous
MeSH Terms: conditions — Peanut Hypersensitivity; Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Viaskin Peanut 250µg (Experimental)
  Interventions: Drug: Viaskin Peanut 250µg

INTERVENTIONS:
Drug: Viaskin Peanut 250µg — DBV712 250 µg, once daily

SUMMARY:
This is an open-label, follow-up study for subjects who completed the PEPITES study. Subjects will be offered enrollment in this follow-up study to receive Viaskin Peanut 250 μg for 2 additional years if previously on active treatment in the PEPITES study, or for 3 years if previously on placebo in the PEPITES study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed the PEPITES study.

Exclusion Criteria:

* Generalized dermatologic disease (for example, active atopic dermatitis, uncontrolled generalized active eczema, ichthyosis vulgaris) extending widely on the skin and especially on the back or arms with no intact zones to apply the Viaskin patches.
* Diagnosis of asthma that evolved to severe, unstable or uncontrolled asthma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2019-11-23 (Actual); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
% of subjects originating from the active arm of PEPITES reaching an Eliciting Dose (ED) ≥ 1,000 mg after 24 months of additional treatment in PEOPLE | Month 24

CONTACTS AND LOCATIONS:
Locations (31):
- United States (17):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of California, Rady Children's Hospital, San Diego, California
  - Stanford University School of Medicine, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Ann & Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Childrens' Hospital, Boston, Massachusetts
  - Jaffe Food Allergy Institute, New York, New York
  - The University of North Carolina - Chapell Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Children's Medical Center of Dallas, Dallas, Texas
  - Baylor College of Medicine - Texas Children's Hospital, Houston, Texas
  - ASTHMA, Inc., Seattle, Washington
- Australia (3):
  - Allergy Medical, Brisbane
  - Princess Margaret Hospital for Children, Perth
  - Children's Hospital Westmead, Sydney
- Canada (6):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Cheema Research Inc., Mississauga, Ontario
  - Ottawa Allergy Asthma Research Institute, Ottawa, Ontario
  - Gordon Sussman Clinical Research Inc., Toronto, Ontario
  - CHUM & CHU Sainte-Justine, Montreal, Quebec
  - Centre de Recherche Appliquée en Allergie de Quebec, Québec
- Germany (3):
  - Charité Universitätsmedizin Berlin, Berlin
  - St.-Marien-Hospital, Bonn
  - Universitätsklinikum Erlangen, Erlangen
- Ireland (2):
  - Clinical Investigations Unit, Cork
  - Our Lady's Children's Hospital, Dublin